CLINICAL TRIAL: NCT04872400
Title: Acute Application Of Intrawound Antibiotic Powder In Open Extremity Fracture Wounds
Brief Title: Acute Application of Antibiotic Powder in Open Fracture Wounds
Acronym: APOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-2957; 5672 (Other Grant/Funding Number: Orthopaedic Trauma Association)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Fractures, Open; Wounds and Injuries--Infections; Anti-Bacterial Agents; Fractures, Bone; Extremity Fracture Lower; Extremity Fractures Upper
Keywords: Open fractures; Antibiotic powder; Vancomycin; Tobramycin; Infection; Gustilo; 16S
MeSH Terms: conditions — Fractures, Open; Wounds and Injuries; Fractures, Bone; Infections | interventions — Vancomycin; Tobramycin

STUDY DESIGN:
Intervention Model Description: The management of open fractures involves an expedited administration of systemic antibiotics and while effective in reducing the rate of infection, complications from infections are still common following open fractures. This trial aims to evaluate the incidence of surgical site infections using topical vancomycin antibiotic powder or topical tobramycin antibiotic powder in combination with standard of care treatment and to evaluate the effectiveness of both topical antibiotic powders in reducing surgical site infection.
Who Masked: Participant
Masking Description: This will be a single-blind study as only the participants will be blinded to the treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects randomized to the Control Arm will receive standard of care open fracture wound care (no powder) by the clinical team.
- Vancomycin (Experimental): Subjects randomized to the Intervention arm will receive standard of care plus 1 gram of vancomycin powder applied topically to the wound bed before the dressing is applied. Intervention will occur in the emergency room prior to surgical intervention.
  Interventions: Drug: Vancomycin
- Tobramycin (Experimental): Subjects randomized to the Intervention arm will receive standard of care plus 1.2 grams of tobramycin powder applied topically to the wound bed before the dressing is applied. Intervention will occur in the emergency room prior to surgical intervention.
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Vancomycin — 1 vial of Vancomycin 1g powder applied topically to the open fracture wound injury.
  Arms: Vancomycin
Drug: Tobramycin — 1 vial of Tobramycin 1.2g powder applied topically to the open fracture wound injury.
  Arms: Tobramycin

SUMMARY:
The purpose of this study is to help determine the best treatment for severe injures like open fracture wounds.

Some broken bone injuries can be more likely to get an infection. It is mostly due to the way they were injured. Surgical site infection in the orthopedic surgery population is a big public health issue. Wound infections result in both longer length of hospital stay and total cost of care. This study will be using an antibiotic called Vancomycin or Tobramycin in a powder form.

DETAILED DESCRIPTION:
The investigators aim to investigate the effectiveness of preoperative intrawound antibiotic powder in preventing infection and reducing bacterial burden after open fracture.

The investigators hypothesize that the participants who receive preoperative intrawound antibiotic powder will have fewer superficial and deep surgical site infections compared to participants who do not receive the antibiotic powder. The investigators also anticipate that the application of the antibiotic powder to open fracture wounds preoperatively will decrease the bacterial burden.

Sample swabs will be analyzed using the 16S metagenomics sequencing on the Illumina platform. Both RNA and DNA extracts will be utilized to identify and quantify the bacterial load in the wound bed at the time immediately prior to surgical debridement.

ELIGIBILITY:
Inclusion Criteria:

* Subject or proxy willing and able to provide written informed consent.
* Age between 18 years and 80 years (inclusive), with an upper or lower extremity Gustilo Type II, IIIA, or IIIB open fractures requiring debridement and internal fixation.
* Open extremity fractures
* Time from injury to study intervention 24 hours or less

Exclusion Criteria:

* Individuals under the age of 18 years or over 80 years
* Type I or IIIC open fractures
* Over 24 hours from time of injury
* Subjects who have received acute operative care of the open fracture at an outside facility prior to presenting at the Emergency Department.
* Open fractures distal to the wrist and midfoot
* History of chronic infection in the extremity involved.
* Subjects who are currently pregnant
* Subjects who are Prisoners
* Subjects with a known allergy to vancomycin or tobramycin
* Subjects with a condition or social circumstances that would reduce adherence and follow-up.
* Subjects Participating in other clinical research involving investigational antimicrobial products within 30 days of randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection during the post-operative follow-up period | Within 6 months of injury date
  The percentage of participants who develop an infection at the surgical site following debridement and fixation at the follow up period.

SECONDARY OUTCOMES:
Shannon's index measure of bacterial diversity based on wound cultures | Within 1 year of injury date
  Characterize species and determine whether changes in biodiversity differ across study arms.
Simpson index measure of bacterial diversity based on the wound cultures | Within 1 year of injury date
  Consider the number of bacterial species present, alongside the relative abundance of each specie across study arms.
Presence of bacterial species commonly attributed to surgical site infections based on would cultures including: Staph, enterococcus, acinetobacter, enterobacter, e. coli, klebsiella, and pseudomonas | Within 1 year of injury date
  Understand the changes that occur in the presence of bacterial species associated with surgical site infection after antibiotic powder treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Alfonso, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No